CLINICAL TRIAL: NCT04843423
Title: An Open-label, Flexible Dose, Single Site Study Evaluating the Safety, Efficacy and Tolerability of Cariprazine as an Adjunct to Psychostimulants in Adult Patients With ADHD Who Have Had an Inadequate Response to Psychostimulants Alone
Brief Title: Adjunct Treatment With Cariprazine for Adults With Attention-deficit/Hyperactivity Disorder
Acronym: ADHD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Martin A. Katzman (Other)
Responsible Party: Sponsor-Investigator, Dr. Martin A. Katzman, Clinic Director, START Clinic for Mood and Anxiety Disorders
Organization: START Clinic for Mood and Anxiety Disorders (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2018-10403
Record Dates: First submitted 2021-03-29; First posted 2021-04-13 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Inattention; Impulsive; Hyperactive; Non-remitting; Treatment resistant
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Impulsive Behavior; Spasm | interventions — cariprazine

STUDY DESIGN:
Intervention Model Description: Longitudinal, open-label, single arm, within-subject, adjective flexible-dose intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cariprazine treatment (Experimental)
  Interventions: Drug: Cariprazine

INTERVENTIONS:
Drug: Cariprazine — At the screening visit, those who are eligible will enter an open-label trial with cariprazine in doses ranging from 1.5mg to 3 mg. The study will begin with a single week of cariprazine 1.5 mg oral tablets. After the first week the participants' dosage may be increased up to a maximum of 3 mg daily. This dose will remain fixed after 4 weeks of treatment until week 8, at which time the medication will be discontinued.
  Because the drug is not yet available to market in Canada, participants will be dispensed the drug in appropriately labelled 7-day tablet containers with the appropriate dose, including 3 additional tablets to account for scheduling conflicts. Participants will be instructed to return the tablet containers at each Study Visit in order to assess drug compliance. They will then be newly dispensed the appropriate quantity according to their next scheduled study visit.

SUMMARY:
According to the Canadian ADHD Practice Guidelines, psychostimulants are the preferred treatment of attention-deficit/hyperactivity disorder (ADHD), especially for those that require urgent care. Specifically, long-acting psychostimulants are considered the gold-standard pharmacological treatment for ADHD. Using extended-release formulations, long-acting psychostimulants provide an extended duration of daily symptom relief in addition to overall reductions in ADHD symptoms that are maintained over time.

In accordance with these guidelines, clinicians may combine psychostimulants with other medications when it is considered necessary. For complex cases, psychostimulants alone are often inadequate for improving the effects of ADHD and are therefore prescribed in conjunction with other medications. At low doses, antipsychotics have been considered appropriate adjunctive medications. Studies show that most adult cases with ADHD that were undiagnosed or untreated in childhood result in the need for adjunctive medication in adulthood to enhance the effects of the psychostimulant. As a result, it is hypothesized that adjunct treatment with a low dose of cariprazine, an atypical antipsychotic, will enhance the effectiveness of standard ADHD treatment with a long-acting psychostimulant in a subset of the ADHD population that achieved little to no response on psychostimulants alone.

DETAILED DESCRIPTION:
According to the Canadian ADHD Practice Guidelines, psychostimulants are the preferred treatment of ADHD, especially for individuals that require urgent care. Specifically, long-acting psychostimulants are considered the first-line pharmacological treatment for ADHD. Utilizing sustained-release mechanisms, long-acting psychostimulants provide an extended duration of daily symptom relief in addition to overall reductions in ADHD symptoms that are maintained over time. Long-acting psychostimulants minimize several of the limitations of immediate-release psychostimulants including: peak-trough effects, suboptimal duration of action, increased diversion potential, and non-adherence due to multiple dosages.

In accordance with these guidelines, clinicians may combine psychostimulants with other medications when it is deemed necessary. For complex cases, psychostimulants alone are often inadequate for ameliorating the debilitating effects of ADHD and are therefore prescribed in conjunction with other psychotropic medications targeted at the residual symptoms associated with ADHD. Antipsychotics have been deemed appropriate as adjunctive medications, especially for the management of reactive-impulsive behaviours, neurological tics, and/or bipolar disorder. Studies show that most adult cases with ADHD that were undiagnosed or untreated in childhood result in the use of adjunctive medication in adulthood to augment the effects of the psychostimulant. As a result, we propose that adjunct treatment with cariprazine, an atypical antipsychotic, will augment the efficacy of standard ADHD treatment with a long-acting psychostimulant in a subset of the population that achieved little to no response on psychostimulants alone.

Cariprazine is an atypical antipsychotic where the active ingredient is cariprazine hydrochloride (HCl). It is a dopamine D3/D2 receptor partial agonist, with a higher affinity for D3 receptors as demonstrated in both in vitro and in vivo studies. It was approved by the FDA in 2015 for the acute treatment of mania/mixed episodes associated with bipolar I disorder in adults and for the treatment of schizophrenia. Its use is also being explored in the treatment of major depressive disorder. Cariprazine capsules are intended for oral administration and should be stored between 20-25 °C. Each hard gelatin capsule contains a white to off-white powder of cariprazine HCl, which is equivalent to either 1.5, 3, 4.5, or 6 mg of cariprazine base.

Overall efficacy and tolerability of cariprazine appears to be good despite some adverse events including akathisia, insomnia, headache, and weight gain. However, most studies reported that the adverse events were mild to moderate. Prior to discussing the mechanism of action of cariprazine and its utility in the present study, we first present a concise review of dopamine transmission and its relevance to ADHD.

Dopamine (DA) neurons are involved in acquisition and reinforcement learning thought to be maintained in part through the mesolimbic dopaminergic system, with projections from the ventral tegmental area (VTA) to regions such as the nucleus accumbens (NAc). The DAergic neurons in the midbrain are the main source of the neurotransmitter (NT) and mediate a wide range of brain functions and behavioural processes such as voluntary movement, mood, reward, addiction, and stress. In addition to the VTA, dopamine neurons expressing D1 and D2 receptors are typically found in the NAc, substantia nigra (SN), striatum, and hippocampus.

The DA neurons exhibit two activity states that mediate separate aspects of behavior. Phasic DA release mainly activates D1 receptors, whereas tonic DA release mainly activates the higher affinity D2 receptors. Phasic activity is thought to facilitate cue-reward acquisition and acquisition of incentive salience, whereas tonic activity is involved in response inhibition and behavioural flexibility. D2 receptor stimulation has been shown to act in opposition to D1 receptors in the regulation of substrates downstream of cyclic adenosine monophosphate (AMP). Furthermore, D2 receptor function appears to play a critical role in the maintenance of reward functions via the NAc as suggested by pharmacological studies. Recent findings also indicate that phasic DA release drives a rapid activation of D2 neurons, suggesting that some of the behavioural effects of phasic release may be partially mediated by D2 signaling.

It has been hypothesized that the D1 pathway is involved in promoting reward responses while the D2 pathway may mediate the opposite response. Phasic DA events are also proposed to indicate the importance of learned reward-predictive cues that drive motivated behavior. Moreover, D3 receptors (D3R), a D2-like receptor, are present in high density in the ventral striatum, which is a cross-section of neural networks involved in processes of reward, motivation, and decision making, and are thought to be tonically occupied by endogenous DA. Due to the projections to/from the prefrontal cortex, abnormal activity at these receptors may be a potential marker for prefrontal deficits, which underlie the comorbidity between ADHD and depression and often contributes to treatment resistance in a subgroup of the population. Cariprazine is therefore assumed to act by exerting antagonist-like actions by inhibiting the binding of the full agonist DA.

Cariprazine was found to be unique among antipsychotics in its ability to increase dopaminergic D3R levels in D3R-rich brain regions following chronic treatment. The exact mechanisms of action underlying cariprazine's effects have not been fully elucidated. Zimnisky et al. (2013) found that in D3R knockout mice, cariprazine demonstrated D3R-dependent protective effects on cognitive function. In addition, Duric et al. (2017) recently reported that cariprazine significantly attenuated chronic unpredictable stress-induced anhedonia-like behaviour in wild-type mice. This effect was not observed in D3R knockout mice, suggesting that the activity is dependent upon D3Rs.

This is significant because alterations in reward circuitry, particularly involving the prefrontal cortex, have been observed in ADHD. Specifically, neurotransmitter studies have revealed abnormalities in DA and norepinephrine (NE) signaling in ADHD. DA and NE activity are associated with many prefrontal cortex functions, including those involved in the attentional control system, reward acquisition and maintenance and maintenance of hedonic tone. Of further interest is the relationship of serotonin (5-HT) to DA and NE because 5-HT is hypothesized to decrease DA and NE activity through 5-HT binding to the 5-HT2a and 5-HT2c receptors respectively. It appears that at lower doses, cariprazine is considered a DA receptor partial agonist, which may serve to increase striatal DA activity, thereby improving aberrant reward system functioning in individuals with ADHD. At higher doses, cariprazine, like most antipsychotics, functions as a DA receptor antagonist, thereby further reducing DA activity. In theory, higher doses of cariprazine should not improve ADHD symptoms.

The DA theory of ADHD states that ADHD results from DA deficits, specifically lowered activity in the frontal cortex and striatum, and is supported by a variety of pharmacological and imaging studies. Given the role of this hypothesized deficit in reward maintenance and specifically in hedonic tone among ADHD patients, adjunctive treatment with low dose cariprazine, a D2/D3R agonist, may have the ability to elevate DA activity in the frontal cortex and ventral striatum and help attenuate dysfunction of the reward circuitry in complex and severe ADHD patients. For the present study, we are particularly interested in the potential action of adjunctive low dose cariprazine in the treatment of ADHD with or without comorbidities for individuals who have had inadequate response to psychostimulants alone. The trial will be conducted in compliance with the protocol, Good Clinical Practice (GCP) guidelines, and with applicable Health Canada regulatory requirements. Site-specific Standard Operating Procedures (SOPs) for conducting clinical trials will be followed for the recruitment of participants, adverse event reporting, and for the collection, management and analysis of data throughout the duration of the study.

Study Population Participants (N = 15) with a primary diagnosis of ADHD using diagnostic and statistical manual of mental disorders (DSM)-5 criteria, with or without comorbid secondary illnesses, who meet all other inclusion/exclusion criteria are eligible for entry into the study. We have chosen to assign 10 potential patients as the number of desired completers (N = 10). Given that the dropout rate with dose adjustment is estimated to be approximately 33 percent, we will enroll a total of 15 participants to complete the study.

All participants will be assigned a participant identification number to maintain patient confidentiality. Binders will be created for each participant using their unique study-specific participant ID in order to store and maintain source documents according to the visit number throughout the duration of the study. Physical binders will be stored in a locked research office at the site. Source documents both related and unrelated to the current study will also be stored electronically in a PHIPA-compliant electronic medical record system. All source documents will be de-identified and will be identifiable only to members of the study personnel through a password-protected document that contains participant names and their corresponding participant IDs. Participant data will be entered into the statistical analysis software (SPSS) using the unique participant IDs in order to maintain patient confidentiality. The study investigator will permit trial-related monitoring, audits, IRB/IEC review, and regulatory inspection(s), providing direct access to source data and documents.

Statistical Plan To evaluate the efficacy of adjunct cariprazine (1.5 - 3 mg, daily) in the treatment of ADHD with or without comorbidities, each participant will act as his/her own control (within-subjects design) and will be evaluated based on pre-treatment and post-treatment responses on the primary and secondary outcome measures. The research question is as follows: Does treatment with adjunct cariprazine improve ADHD symptoms in participants that are on a stable dose of their psychostimulant who have not yet achieved remission? H0 Adjunct treatment with cariprazine does not improve ADHD symptoms. H1 Adjunct treatment with cariprazine improves symptoms of ADHD in outpatients who are on a stable dose of an existing psychostimulant and have not yet achieved remission.

To answer the research question, a within-subjects t-test will be performed to compare baseline and post-treatment total scores on the primary ADHD measure.

Secondary analyses will employ a series of within-subjects t-tests to evaluate the relationship between cognition, energy and motivation, and hedonic tone at baseline compared to post-treatment of 8 weeks with adjunct cariprazine. There are no plans for interim analysis at this time. No pharmacokinetic analyses will be undertaken.

Response or remission on the primary ADHD outcome measure will be assessed, in addition to statistical analyses testing significance of absolute change in total scores. All parametric tests will be 2-tailed and performed at a 5 percent alpha level. Descriptive statistics will be provided by assessments for the total score and changes from baseline in the total score on all of the measures used. Data based on observed cases and last observation carried forward will be summarized. Overall, the safety and tolerability of cariprazine in participants with ADHD will be assessed by changes from baseline in physical examination, clinical laboratory test results, and vital signs. Safety analyses will be presented by means of descriptive statistics, frequency tables and graphical presentations as appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. The participant has provided signed informed consent.
2. Males and/or females aged 18-70 (extremes included).
3. Participants with a primary diagnosis of ADHD according to DSM-5 (314.01) criteria (diagnosis to be made using the Mini-International Neuropsychiatric Interview (MINI) 7.0.2 and confirmed by the Diagnostic Interview for ADHD in Adults (DIVA 5.0). Participants with a comorbid anxiety and depressive disorder will be permitted, as long as ADHD is judged to be the primary diagnosis.
4. Participants who score an ASRS of ≥ 4 in Part A at both Screening and Baseline, representing non-response to current stable psychostimulant treatment
5. Participants are on a stable dose (> 4 weeks) of their existing long-acting psychostimulant (any type) prior to entry into the study.
6. Participants are on a stable dose of any other psychotropic medication (> 8 weeks) to treat comorbid conditions, except antipsychotics.
7. On the basis of a physical examination, medical history and basic laboratory screening, the patient is, in the investigator's opinion, in a suitable condition.

   Basic laboratory screening includes:

   Chemistry: Electrolytes, ALT, Albumin, Alkaline Phosphatase, AST, Bilirubin Total protein, Creatinine, Urea (BUN), CK, GGT, Potassium, Sodium, Calcium, Glucose (Fasting), Bilirubin Direct, Bicarbonate, Chloride, Urate (for Uric Acid), LD, Magnesium, Phosphorus, Amylase CBC: Hematocrit, Hemoglobin, RBC, WBC + differential, abs. Platelet Count Drug Screen (urine-8 tests): amphetamines, benzodiazepines, barbiturates, methadone, cocaine, opiates, cannabinoids, PCP Standard Urinalysis Lipid Assessment: Cholesterol, HDL, LDL-calc, Triglycerides Prolactin
8. Willing and able to attend study appointments in the correct time windows.

Exclusion Criteria:

Participants meeting one or more of the following criteria cannot be selected for inclusion:

1. Any other primary mental health disorder in the previous six months.
2. Alcohol or drug abuse as defined in the DSM-5 criteria within the last six months.
3. Mania, hypomania as defined in the DSM-5 criteria.
4. Any psychotic disorder.
5. Eating disorders as defined in the DSM-5 criteria.
6. Any cognitive disorder or dementia within 3 months before the baseline visit.
7. A history of Seizure Disorder (Epilepsy or other).
8. Clinical interpretation of apparent suicide risk.
9. Commencement of formal psychotherapy for 4 weeks prior to entry into the study and/or during the course of the study.
10. Existing treatment with any antipsychotic as mono- or adjunct therapy at the time of the study.
11. Change in use of medications.
12. Laboratory values at screening or in medical history that may be considered through clinical interpretation to be significant, including positive drug and alcohol tests.
13. Diseases that could through clinical interpretation interfere with the assessments of safety, tolerability and efficacy of study treatment.
14. Serious illness: liver or renal insufficiency, cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurological, infectious, neoplastic or metabolic disturbance.
15. If female, the subject is pregnant or lactating or intending to become pregnant before, during, or within 30 days after participating in this study, or intending to donate ova during such time period.
16. The participant has received electroconvulsive therapy, vagal nerve stimulation, or repetitive transcranial magnetic stimulation within 6 months prior to Screening.
17. The participant is, in the opinion of the investigator, unlikely to be able to comply with the clinical trial protocol or is unsuitable for any other reasons.
18. Contraindications and Warning Precautions as per the U.S. Product Monograph will be followed.

Participants must discontinue the use of recreational drugs including cannabis for at least 2 weeks prior to entry into the study. Participants must limit alcohol intake to a maximum of 3 standard drinks per week during the study period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-04-14 (Estimated)

PRIMARY OUTCOMES:
Mean changes in the ADHD Rating Scale (ADHD RS-5) | Pre treatment (screening, week 0) and post treatment (week 8)
  Remission cut off score is defined as less than or equal to 18

SECONDARY OUTCOMES:
Mean changes on the Barkley Adult ADHD Rating Scale IV (BAARS-IV) | Pre treatment (screening, week 0) and post treatment (week 8)
  Where response rate is defined at 50 percent improvement in symptoms
Mean changes on the Adult ADHD Self-Report Scale (ASRS) v1.1 | Pre treatment (screening, week 0) and post treatment (week 8)
  Where remission is greater than 14
Mean changes on the Intolerance of Uncertainty Scale (IUS) | Pre treatment (screening, week 0) and post treatment (week 8)
  self-report measure of intolerance of uncertainty, where lower scores indicate greater capacity to tolerate ambiguity
Mean changes on the Clinical Global Impression - Severity (CGI-S) scale | Pre treatment (screening, week 0) and post treatment (week 8)
  where response rate is measured as 50 percent improvement on the CGI-S
Mean changes in on the Time Sensitive ADHD Symptom Scale (TASS) | Pre treatment (screening, week 0) and post treatment (week 8)
  self-report inventory assessing severity of ADHD symptoms throughout the day
Mean changes on the Fawcett-Clark Pleasure Capacity Scale (FCPS) | Pre treatment (screening, week 0) and post treatment (week 8)
  Self-report inventory assessing anhedonia or hedonic tone
Mean changes on the cognitive battery | Pre treatment (screening, week 0) and post treatment (week 8)
  Cambridge Health Sciences neuropsychological assessment battery including memory, reasoning, verbal ability, and concentration tasks
Mean changes on the Snaith-Hamilton Pleasure Scale (SHAPS) | Pre treatment (screening, week 0) and post treatment (week 8)
  Self-report inventory assessing anhedonia or hedonic tone
Mean changes on the Dimensional Anhedonia Rating Scale (DARS) | Pre treatment (screening, week 0) and post treatment (week 8)
  Self-report inventory assessing anhedonia
Mean changes on the Motivation and Energy Inventory (MEI) | Pre treatment (screening, week 0) and post treatment (week 8)
  self-report inventory assessing motivation and energy as a proxy measure for hedonic capacity

CONTACTS AND LOCATIONS:
Overall Officials: Martin A Katzman, MD, Principal Investigator — Clinic Director
Locations (1):
- START Clinic for Mood and Anxiety Disorders, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No